CLINICAL TRIAL: NCT03927131
Title: Double-blind, Randomized Clinical Trial With Active Controls to Assess Safety, Immunogenicity and Lot-to-lot Consistency of Inactivated Split-virion Quadrivalent Influenza Vaccine of Butantan Institute
Brief Title: Safety and Immunogenicity of the Butantan Quadrivalent Influenza Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Butantan Institute (Other Government)
Collaborators: Butantan Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FLQ-01-IB
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Influenza, Human
Keywords: Vaccines
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- QIV-IB (Experimental): Inactivated split-virion quadrivalent influenza vaccine
  Interventions: Biological: QIV-IB
- TIVV-IB (Active Comparator): Inactivated split-virion trivalent Influenza Vaccine containing Influenza B virus - Victoria lineage
  Interventions: Biological: TIVV-IB
- TIVY-IB (Active Comparator): Inactivated split-virion trivalent Influenza Vaccine containing Influenza B virus - Yamagata lineage
  Interventions: Biological: TIVY-IB
- QIV-IB Lot A (Experimental): Inactivated split-virion quadrivalent influenza vaccine - Lot A
  Interventions: Biological: QIV-IB Lot A
- QIV-IB Lot B (Experimental): Inactivated split-virion quadrivalent influenza vaccine - Lot B
  Interventions: Biological: QIV-IB Lot B
- QIV-IB Lot C (Experimental): Inactivated split-virion quadrivalent influenza vaccine - Lot C
  Interventions: Biological: QIV-IB Lot C

INTERVENTIONS:
Biological: QIV-IB — Inactivated split-virion quadrivalent influenza vaccine
  Arms: QIV-IB
Biological: TIVV-IB — Inactivated split-virion trivalent Influenza Vaccine containing Influenza B virus - Victoria lineage
  Arms: TIVV-IB
Biological: TIVY-IB — Inactivated split-virion trivalent Influenza Vaccine containing Influenza B virus - Yamagata lineage
  Arms: TIVY-IB
Biological: QIV-IB Lot A — Inactivated split-virion quadrivalent influenza vaccine - Lot A
  Arms: QIV-IB Lot A
Biological: QIV-IB Lot B — Inactivated split-virion quadrivalent influenza vaccine - Lot B
  Arms: QIV-IB Lot B
Biological: QIV-IB Lot C — Inactivated split-virion quadrivalent influenza vaccine - Lot C
  Arms: QIV-IB Lot C

SUMMARY:
Studies have shown that a broader spectrum influenza vaccine may help in reducing the influenza burden of disease. Butantan Institute is currently developing a quadrivalent influenza vaccine candidate. This study is will provide safety and immunogenicity data on this quadrivalent influenza vaccine candidate.

The study will be conducted in an open population of healthy participants (3 years old and above) recruited in different clinical sites in Brazil and will be adequately powered to assess safety, immune response (measured by GMT HI antibodies) to each viral strain in the vaccines and lot-to-lot consistency.

DETAILED DESCRIPTION:
This is a double blinded, randomized active-control comparator study to assess the safety and immunogenicity of QIV-IB, the Butantan Institute quadrivalent influenza vaccine candidate. As active controls, two trivalent influenza vaccines with different Influenza B strains, one with influenza B/Victoria strain (TIVV-IB) and other with influenza B/Yamagata strain (TIVY-IB).

The study is designed to build a safety database of the quadrivalent influenza vaccine in adults to detect adverse events with a frequency of 1:1000 or higher and safety databases for elderly and pediatric age groups to detect adverse events with frequency of 1:100 or higher.

In terms of immune response, the study aims to demonstrate superiority of HI (Hemagglutinin inhibition) GMT (Geometric Mean Titer) of the QIV-IB for the Influenza B strain that is not present in each trivalent vaccine control. Regarding the Influenza A and B strains common to QIV-IB and both trivalent vaccine controls, the study aims to demonstrate non-inferiority on those strains.

Finally, a lot-to-lot consistency test will be performed in a sub-group of adult participants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 3 years or older at the time of enrollment.
* Provide written informed consent
* Agrees to complete all study visits, procedures and contacts
* Women and adolescents of childbearing age: Negative pregnancy test with understanding (through informed consent process).

Exclusion Criteria:

* Chronic medical conditions such as psychiatric conditions, diabetes, hypertension or any other conditions that might place the subjects at high risk of adverse events. Study clinicians will use clinical judgment on a case-by-case basis to assess safety risks under this criterion.
* Clinically significant abnormalities on physical examination.
* Use of immunosuppressive medications such as systemic corticosteroids or chemotherapeutics, or immunosuppressive illness.
* Women who are pregnant or planning to become pregnant during the study period plus 3 months beyond the last vaccine dose and currently nursing women.
* Participation in research involving another investigational product within 30 days before planned date of first vaccination or anytime through the last study safety visit.
* Clinically significant abnormalities on basic laboratory screening tests.
* Acute febrile illness (axillar temperature ≥ 37.8°C)
* Hypersensitivity to egg or chicken proteins or any of the vaccine constituents
* Thrombocytopenia or a bleeding disorder contraindicating intramuscular vaccination
* Unstable chronic illness (defined as illness requiring hospitalization or a clinically significant change in medication in the previous 12 weeks).
* Alcohol abuse of alcohol or drug addiction
* Any vaccination within the previous 4 weeks
* Seasonal influenza vaccination in the current year

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 5822 (Actual)
Dates: Start 2021-05-12 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2024-03-13 (Actual)

PRIMARY OUTCOMES:
Safety through number of Adverse Events of QIV-IB, TIVV-IB, TIVY-IB per age group | 07 days post-vaccination
  Frequency and intensity of solicited and unsolicited adverse reactions
Safety through number of Adverse Events of QIV-IB, TIVV-IB, TIVY-IB per age group | 42 days post-vaccination
  Frequency and intensity of unsolicited adverse reactions and adverse events of special interest
Superiority for influenza B/Victoria strain | 21 days post-vaccination
  HI GMT ratio for Influenza B/Victoria strains between QIV-IB and TIVY-IB
Superiority for influenza B/Yamagata strain | 21 days post-vaccination
  HI GMT ratio for Influenza B/Yamagata strains between QIV-IB and TIVV-IB
Non-inferiority for common influenza strains between QIV-IB, TIVV-IB and TIVY-IB | 21 days post-vaccination
  HI GMT ratios for Influenza strains between QIV-IB, TIVV-IB and TIVY-IB
Lot-to-lot consistency for immune response to different lots of QIV-IB | 21 days post-vaccination
  HI GMT ratios for Influenza among QIV-IB strains towards among of different lots (A, B and C)

CONTACTS AND LOCATIONS:
Overall Officials: Fernanda Castro Boulos, MD, Study Director — Instituto Butantan
Locations (12):
- Brazil (12):
  - Centro de Pesquisa Clínica Universidade Federal do Ceará - UFC (Site FOR01), Fortaleza, Ceará
  - Núcleo de Pesquisa e Desenvolvimento de Medicamentos - NPDM - Universidade Federal do Ceará - UFC (Site FOR 01), Fortaleza, Ceará
  - Centro de Pesquisa e desenvolvimento de fármacos (Site BHZ01), Belo Horizonte, Minas Gerais
  - Centro de Pesquisa Clínica Real Hospital Português de Beneficência em Pernambuco (Site REC01), Recife, Pernambuco
  - Centro de Pesquisa Clínica Hospital Escola da Universidade Federal de Pelotas (Site PET01), Pelotas, Rio Grande do Sul
  - Centro de Pesquisa Clínica do Hospital São Lucas da PUCRS (Site POA01), Porto Alegre, Rio Grande do Sul
  - Centro de Pesquisas Clínicas da Universidade Federal de Sergipe (Site AJU01), Laranjeiras, Sergipe
  - Centro de Pesquisa Clínica Faculdade de Medicina de Ribeirão Preto da Universidade de São Paulo (FMRPUSP) (Site RAO01), Ribeirão Preto, São Paulo
  - Centro de Pesquisa Clínica da Universidade Municipal de São Caetano do Sul (Site SCS01), São Caetano do Sul, São Paulo
  - Centro de Pesquisa Clínica Fundação Faculdade Regional de Medicina de São José do Rio Preto (Site SJP01), São José do Rio Preto, São Paulo
  - Centro de Pesquisa Clínica Serrana (Site RAO03), Serrana, São Paulo
  - Centro de Pesquisas Clínicas do Instituto Central da FMUSP Unidade II (Site SAO01), São Paulo

IPD SHARING:
Plan to Share IPD: No